CLINICAL TRIAL: NCT05943197
Title: Clinical and Microbiological Approach in Orthopedic Treatment of Patients When Choosing a Structural Material
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samara State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/2022
Record Dates: First submitted 2023-02-25; First posted 2023-07-13 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Oral Microbiota
Keywords: microbiota
MeSH Terms: interventions — Microbiota

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 20 patients with zirconia (Experimental): patients who will receive crowns from zirconia
  Interventions: Diagnostic Test: dental prosthetics, biofilm response and oral microbiota
- 20 e-max patients (Experimental): patients who will receive crowns from e-max
  Interventions: Diagnostic Test: dental prosthetics, biofilm response and oral microbiota
- 20 patients Cobalt-chromium alloy (Experimental): patients who will receive crowns from Cobalt-chromium alloy
  Interventions: Diagnostic Test: dental prosthetics, biofilm response and oral microbiota
- 20 patients metal-ceramics (Experimental): patients who will receive crowns from metal-ceramics
  Interventions: Diagnostic Test: dental prosthetics, biofilm response and oral microbiota

INTERVENTIONS:
Diagnostic Test: dental prosthetics, biofilm response and oral microbiota — microbiota, biofilm, oral mucosa

SUMMARY:
Today, there is a wide range of structural materials on the market, different in chemical, physical and biological properties, and information about them is very often limited only by the manufacturer's instructions, which allows to determine, at best, only the scope. In this regard, there are difficulties in choosing the optimal material for this particular situation, since without a thorough approach to studying the properties of the main materials used in dentistry, it seems difficult to provide high-quality dental care, the result of which is functional usefulness, aesthetics and durability.The problem of an individual approach to the choice of structural material from the standpoint of personalized medicine is even less studied - there are no data in the literature on the role of normal and pathogenic microflora in the development of destructive changes in structures and the development of complications, taking into account a personalized approach when analyzing the composition of the microbiota of the oral cavity, biochemical parameters of the oral fluid, blood depending on the material from which the structure is made.

DETAILED DESCRIPTION:
Relevance of the topic Today, there is a wide range of structural materials on the market, different in chemical, physical and biological properties, and information about them is very often limited only by the manufacturer's instructions, which allows to determine, at best, only the scope. In this regard, there are difficulties in choosing the optimal material for this particular situation, since without a thorough approach to studying the properties of the main materials used in dentistry, it seems difficult to provide high-quality dental care, the result of which is functional usefulness, aesthetics and durability.The problem of an individual approach to the choice of structural material from the standpoint of personalized medicine is even less studied - there are no data in the literature on the role of normal and pathogenic microflora in the development of destructive changes in structures and the development of complications, taking into account a personalized approach when analyzing the composition of the microbiota of the oral cavity, biochemical parameters of the oral fluid, blood depending on the material from which the structure is made.

Purpose of the study Improving the efficiency of orthopedic treatment of patients with dentition defects based on a clinical and microbiological personalized approach

Research objectives:

1. Conduct an analysis of the need for fixed orthopedic structures among the population at the regional level
2. Assess the influence of the material chosen for prosthetics on the species diversity of oral microorganisms
3. To study the dependence of the degree of microbial adhesion on the nature of the material and manufacturing technology on various fixed orthopedic structures
4. Develop and implement a method for preventing complications in patients with prosthetics using various structural materials
5. Conduct a comparative assessment of the orthopedic treatment of patients using the developed method for the prevention of complications and the traditional method based on clinical and functional research methods

Material (object) of research:

The clinical part of the study is carried out at the Department of Orthopedic of dentistry of Samara State Medical University on the basis of GBUZ SO SSP No. 3 g.o. Samara. To solve the tasks of the study, an analysis of the clinical observation of patients. Planned orthopedic treatment 20 patients with zirconia 20 e-max patients 20 patients Cobalt-chromium alloy 20 patients Biological material will be taken from each patient before the delivered structure and after 1 month of the structure's arrival in the oral cavity

Research methods:

Clinical

* hygiene indexes
* CPU index Microbiological
* MALDI-ToF mass spectrometry Clinical diagnostic research
* biochemical study of saliva
* biochemical blood test X-ray examination Scientific novelty of the work

  1. For the first time, a personalized approach will be developed in the choice of structural material for the manufacture of dentures based on a clinical and microbiological study
  2. For the first time, an analysis of the results of treatment and the development of complications will be carried out using the proposed method.
  3. For the first time, a cultural study of the composition of microorganisms of the oral mucosa will be carried out, depending on the selected material
  4. For the first time, a model of microbiological examination of patients will be scientifically substantiated when choosing a structural material Practical significance

     * For the first time, an algorithm for orthopedic treatment will be proposed when choosing a structural material depending on the microbiology of the oral cavity
     * For the first time, methods will be proposed for determining the influence of oral microflora on orthopedic structures, taking into account individual characteristics
     * For the first time, an algorithm for microbiological examination of patients for prosthetics will be proposed
     * For the first time, biomarkers will be proposed to assess the microbial composition of the oral cavity to justify the choice of design

ELIGIBILITY:
Inclusion Criteria:

- need for prosthetics

Exclusion Criteria:

- lack of indications for treatment

Ages: 1 Month to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
microbiological research | 1 month after placing a crown in the mouth
  Before the installation of an orthopedic structure in the oral cavity, microbiological material is taken from the periodontal cavity of the tooth on which the orthopedic structure will be installed. Next, an orthopedic structure is installed for a period of 1 month, after which the structure is removed from the oral cavity, for re-analysis and comparison of changes in the microbiota of the oral cavity, depending on the selected structural material There will be measurements of the size of the tissues of the oral cavity, depending on the choice of material for prosthetics, using molecular genetic, biochemical, microbiological studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Gbuz So Sspn3, Samara, Russia

IPD SHARING:
Plan to Share IPD: No